CLINICAL TRIAL: NCT06560294
Title: Glue Embolization Versus Conservative Treatment for Pelvic Congestion Syndrome: A Randomized Trial
Brief Title: Glue Embolization vs Conservative Treatment for Pelvic Congestion Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Adel Eleissawy, Lecturer of Vascular and Endovascular Surgery, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR752/7/24
Record Dates: First submitted 2024-08-11; First posted 2024-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Glue Embolization; Pelvic Congestion Syndrome
MeSH Terms: interventions — Diosmin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micronized purified flavonoid fraction (Daflon ®) (Active Comparator): Patients will receive micronized purified flavonoid fraction (Daflon ®), 500 mg twice/daily for 3 months.
  Interventions: Drug: Micronized purified flavonoid fraction (Daflon ®)
- Glue embolization (Experimental): Patients will receive transcatheter glue embolization.
  Interventions: Other: Glue embolization

INTERVENTIONS:
Drug: Micronized purified flavonoid fraction (Daflon ®) — Patients will receive micronized purified flavonoid fraction (Daflon ®), 500 mg twice/daily for 3 months.
  Arms: Micronized purified flavonoid fraction (Daflon ®)
Other: Glue embolization — Patients will receive transcatheter glue embolization.
  Arms: Glue embolization

SUMMARY:
The aim of this study is to compare glue embolization and conservative treatment for pelvic congestion syndrome regarding safety and efficacy.

DETAILED DESCRIPTION:
Pelvic congestion syndrome (PCS) is a common cause of chronic lower abdominal/pelvic pain, estimated to affect about 40 % of women, predominantly between the ages of 30 and 45.The treatment of PCS depends mainly on the severity of the pain. Non-steroid anti-inflammatory drugs are often used, and contraceptives have a role in cases of pain associated predominantly with menstruation.

Traditionally, conservative approaches, such as pharmacotherapy with venoactive drugs like micronized purified flavonoid fraction (Daflon), have been utilized to address the symptoms of PCS. Daflon has been used to treat venous insufficiency and has demonstrated efficacy in reducing symptoms and improving the quality of life in patients with PCS. Its mechanism of action includes improving venous tone, reducing venous stasis, and exerting anti-inflammatory effects. Endovascular treatment of PCS is challenging and requires occlusion of incompetent pelvic veins.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 30 to 50 years.
* Complaining from pelvic congestion syndrome.

Exclusion Criteria:

* Pregnant women at any gestational age, women who gave birth less than 12 months ago, and breastfeeding mothers.
* Patients who are treated with opiates to reduce pelvic pain in the period before the study.
* Patient with history of contrast allergy
* Patient with renal impairment
* Patient has alternative gynecological cause of chronic pelvic pain as pelvic inflammatory disease (PID), endometriosis, fibroid, adenomyosis, ovarian cyst
* Patient underwent any previous intervention for pelvic congestion syndrome as laparoscopy or surgery.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with pelvic congestion syndrome
Enrollment: 40 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | Post intervention for 3 months
  Degree of pain will be assessed using a Visual Analog Scale (VAS). The VAS is a self-reported scale consisting of a horizontal or vertical line, usually 10 cm long. An introductory question asks the patient to mark a point on the line that best refers to his or her pain. Patients will be encouraged to assess the intensity of subjective manifestation of each symptom by scoring from 0 (no symptom) to 10 (the most extreme manifestation possible).

SECONDARY OUTCOMES:
Incidence of recurrence of pain | Post intervention for 3 months
  Incidence of recurrence of pain will be recorded.
Pelvic Venous Clinical Severity Score (PVCSS) | Post intervention for 3 months
  Assessment of treatment outcomes will be standardized using the disease-specific Pelvic Venous Clinical Severity Score (PVCSS) for female patients with pelvic congestion syndrome. The PVCSS takes into account 10 major symptoms and signs of the disease, each of which is scored from 0 (no symptom) to 3 (maximum severity) for a maximum score of 30, which indicates an extremely severe degree of disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.